CLINICAL TRIAL: NCT04137549
Title: Registry Study on "Control Nocturnal Hypertension to Reach the Target "（CONTROL-NHT）
Brief Title: Registry Study on "Control Nocturnal Hypertension to Reach the Target "
Acronym: CONTROL-NHT
Status: Recruiting | Type: Observational
Sponsor: Shanghai Institute of Hypertension (Other)
Responsible Party: Principal Investigator, Yan Li, Professor of Cardiovascular Medicine, Shanghai Institute of Hypertension
Other Study IDs: CONTROL-NHT
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Nocturnal Hypertension
Keywords: ambulatory blood pressure monitoring; nocturnal hypertension; cardiovascular risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Nocturnal controlled hypertension: Nocturnal blood pressure was controlled under 120/70 mmHg after aggressive anti-hypertensive therapy.
- Nocturnal uncontrolled hypertension: Nocturnal blood pressure was still over 120/70 mmHg after aggressive anti-hypertensive therapy.

SUMMARY:
Ambulatory blood pressure monitoring (ABPM) is a major innovation in the history of hypertension diagnosis. In clinical practice, the most well established indication for using ABPM is to identify patients who have high BP readings in the office but normal readings during usual daily activities outside of this setting or vice versa, and to identify varying 24-h BP profiles. However, in recent years, there has been increasing interest in BP values during sleep, and nocturnal BP is now recognized to be superior to daytime BP in predicting fatal and nonfatal cardiovascular events (stroke, myocardial infarction, and cardiovascular death), especially in medicated patients.

The current direction in the management of hypertension is toward earlier and lower BP control for 24 hours, including the nocturnal and morning periods. Therefore, it may be of great significance to pay attention to the management of nocturnal blood pressure so as to reduce the increased cardiovascular risks.

Information of nocturnal hypertensive patients defined by ABPM was prospectively registered nationwide, and then to investigate whether there was difference in cardiovascular prognosis according to the control of ambulatory nocturnal blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-79 years old
* Clinical diagnosed hypertension with the use of antihypertensive drugs
* Nocturnal hypertension ( nocturnal systolic blood pressure ≥ 130 mmHg and/or nocturnal diastolic blood pressure ≥ 80 mmHg)
* A 24-hour ambulatory blood pressure monitoring was performed with validated equipment.
* Willing to provide information about disease history and blood biochemical test data within 6 months.
* Sign the informed consent

Exclusion Criteria:

* Without antihypertensive drug use
* Hospitalized hypertension patients
* Non-compliant patient

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic, and community sample
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence time of fatal and non-fatal cardiovascular events. | From date of enrollment until date of first documented event assessed up to 3 years
  Fatal and non-fatal cardiovascular events, including cardiovascular mortality, non-fatal myocardial infarction, non-fatal stroke, coronary artery bypass grafting or interventional stenting or balloon dilation, and hospitalization for heart failure.

SECONDARY OUTCOMES:
The occurrence time of all-cause mortality. | From date of enrollment until date of first documented event, assessed up to 3 years
The occurrence time of fatal and nonfatal stroke. | From date of enrollment until date of first documented event assessed up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No